## Official Title

A non-randomized, open-label study to evaluate the safety and effectiveness of Koya active wearable compression technology for treating lower limb lymphedema

NCT Number: NCT04897035

**Protocol Number: KCT 006** 

**Document Date: 01/01/2021** 

| Study Title | A non-randomized, open-label study to evaluate the safety and effectiveness of Koya active wearable compression technology for treating lower limb lymphedema |
|---|---|
| Study Objective | To demonstrate that the Koya active wearable compression technology is safe and effective for use |
| Clinical<br>Hypothesis | 1. The Koya wearable device improves quality of life (LYMQOL®) in subjects with lower extremity edema as measured by the difference between preuse and post-use of the device |
| | 2. The Koya wearable device is safe for use as assessed by adverse events |
| | 3. The Koya active wearable compression device maintains or reduces swelling in patients with lower extremity edema as measured by the difference between pre-use and post-use of the device |
| Subject<br>Population | Up to 50 subjects will be enrolled. |
| Investigational<br>Materials | <ul> <li>The Koya wearable device is a smart calibrated active gradient pressure full-leg compression garment that is segmental and programmable, and applies controlled sequential pressure from the distal to proximal-end of the limb in a cyclic manner. These patterns are similar to advanced pneumatic compression devices, which are known to produce safe, well-regulated compression.</li> <li>A controller with a rechargeable battery that powers the limb garment</li> </ul> |
| Study Design | |
| Structure | Non-randomized, open-label pilot study |
| Number of Sites | Up to six (6) sites. |
| Duration | The duration of subject participation is approximately four (4) months |
| Control | None |
| Visit Schedule | Subjects will be seen at the screening visit, day 0, day 7, and week 4, week 8 and week 12 |
| Clinical | LYMQOL Survey Index |
| Parameters | <ul> <li>Sequential Circumference using Tape Measure</li> <li>Photography of the lower limb</li> </ul> |
| Primary Endpoints | <ul> <li>Photography of the lower limb</li> <li>LYMQOL Index</li> </ul> |
| Secondary | Lower Limb Volume |
| Endpoints | Adverse Event |
| | Adherence (exploratory) |
| Key Inclusion Criteria (not a complete list) | <ul> <li>Males and females ≥ 18 years of age</li> <li>Willing to sign the informed consent and deemed capable of following the study protocol</li> </ul> |
| | <ul> <li>Subjects must have a diagnosis of primary or secondary unilateral lower<br/>extremity edema</li> </ul> |

| • | At the time of initial evaluation, individuals must be at least 3 months |
|---|--------------------------------------------------------------------------|
| | post surgery, chemotherapy and/or radiation treatment for cancer if |
| | applicable. |

## Key Exclusion Criteria (not a complete list)

- Individuals with a history or presence of a systemic disorder or condition that could place the subject at increased risk from sequential compression therapy
- Inability or unwillingness to participate in all aspects of study protocol and/or inability to provide informed consent
- Subjects with exam results that would prevent safe and effective use of the study device (cellulitis, open-wounds, healing-wounds, etc.)
- Subjects must not have any diagnosed cognitive or physical impairment that would interfere with use of the device
- Diagnosis of lipedema
- Diagnosis of active or recurrent cancer (< 3 months since completion of chemotherapy, radiation therapy or primary surgery for the cancer)
- Diagnosis of Acute infection (in the last four weeks)
- Diagnosis of acute thrombophlebitis (in last 6 months)
- Diagnosis of pulmonary embolism or deep vein thrombosis within the previous 6 months
- Diagnosis of pulmonary edema
- Diagnosis of congestive heart failure (uncontrolled)
- Diagnosis of chronic kidney disease with acute renal failure
- Diagnosis of epilepsy
- Subjects with poorly controlled asthma
- Any condition where increased venous and lymphatic return is undesirable
- Women who are pregnant, planning a pregnancy or nursing at study entry
- Participation in any clinical trial of an investigational substance or device during the past 30 days